CLINICAL TRIAL: NCT06008678
Title: A Multicenter, Single-Arm, Safety and Efficacy Study of the Resvent RXiBreeze™ PAP System to Treat Obstructive Sleep Apnea
Brief Title: Study of the Resvent RXiBreeze™ PAP System to Treat Obstructive Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Resvent Holding USA LTD (Industry)
Collaborators: Avania (Industry); Resvent Medical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Resvent Medical Technology Co., Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KF-0611-6-0599
Record Dates: First submitted 2023-08-11; First posted 2023-08-23 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Obstructive Sleep Apnea
Keywords: obstructive sleep apnea; sleep apnea; CPAP; PAP; APAP
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes

STUDY DESIGN:
Intervention Model Description: single-arm trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Treatment (Other): RXiBreeze PAP System, Model RXiBreeze 20A
  Interventions: Device: RXiBreeze PAP System, Model RXiBreeze 20A

INTERVENTIONS:
Device: RXiBreeze PAP System, Model RXiBreeze 20A — The RXiBreeze PAP System is a prescription-only positive airway pressure (PAP) ventilator used to treat obstructive sleep apnea (OSA). It is a microprocessor-controlled device that provides mechanical ventilation to a subject.

SUMMARY:
The goal of this clinical trial is to test the automatic positive airway pressure (APAP) function of the RXiBreeze PAP System in adult subjects with obstructive sleep apnea (OSA). The main questions the study aims to answer are:

1. Is apnea-hypopnea index (AHI) detection using the RXiBreeze PAP System equivalent to apnea-hypopnea index (AHI) detection using PSG?
2. What is the responder rate using the RXiBreeze PAP System?

Participants will use the APAP function of the RXiBreeze PAP System while undergoing polysomnography (PSG) for two separate nights in a sleep center. During each visit, participants will also complete two patient reported outcome questionnaires:

* Epworth Sleepiness Score (ESS); and
* Functional Outcomes of Sleep Questionnaire (FOSQ) short form.

DETAILED DESCRIPTION:
This is a prospective, multicenter, single-arm trial designed to evaluate the safety and effectiveness of the RXiBreeze PAP System to treat obstructive sleep apnea and detect breathing events. Eligible subjects who meet all inclusion criteria and none of the exclusion criteria will be consented for study participation. The study will enroll up to 68 subjects. Baseline PSG will be obtained. Subjects will return to the sleep lab and use the RXiBreeze PAP System while undergoing a PSG. The data from both the RXiBreeze PAP System and PSG from both nights will be sent to an independent core lab for blinded AHI scoring. Data will be evaluated in accordance with current American Academy of Sleep Medicine (AASM) scoring guidelines. In addition to the device/PSG data scoring, subjects will complete the Epworth Sleepiness Score (ESS) and the Functional Outcomes of Sleep Questionnaire (FOSQ) short form (10 questions) and be assessed for device- and/or therapy-related adverse events (AEs) at the end of each visit.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥ 22 years old
2. Subject has been diagnosed with OSA (as scored per AASM scoring guidelines) and has an AHI ≥ 10, based on the results of a sleep study conducted at an accredited sleep lab, within 30 days prior to enrollment
3. Subject weighs >30 kg
4. Subject has been prescribed the use of an Auto CPAP system
5. Subject agrees to fulfill all study-required tests, sleep lab session attendance, and assessments
6. Subject agrees to use the RXiBreeze PAP System as prescribed
7. Subject is willing and able to provide informed consent

Exclusion Criteria:

1. Subject has been diagnosed with a sleep disorder other than OSA
2. Subject's Central Apnea Index from the baseline PSG is > 20% of AHI
3. Subject has been diagnosed with severe (stage 3) coronary artery disease
4. Subject has been diagnosed with bullous lung disease
5. subject has been diagnosed with hypotension
6. subject has been diagnosed with bypassed upper airway pneumothorax
7. Subject is pregnant, breastfeeding, or planning on becoming pregnant during trial participation
8. Subject, in the opinion of the investigator, is not suitable for trial participation

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2023-08-22 (Actual); Primary Completion 2023-11-22 (Actual); Study Completion 2023-11-29 (Actual)

PRIMARY OUTCOMES:
AHI Event Detection | Night 1
  Apnea-Hypopnea Index (AHI) as measured by the test device (RXiBreeze PAP System) will be compared to the AHI as measured by polysomnography (PSG) to determine equivalence at night 1. Equivalence will be considered if the mean difference in detected AHI is greater than the lower equivalence limit (EL) of -5 and less than the upper equivalence limit (EU) of 5.
Responder Rate | Night 1
  RXiBreeze PAP System Night 1 responder rate as compared to a performance goal of 50. Responder rate is based on Sher's Criteria, which are defined as having both a ≥ 50% reduction in AHI and a final AHI of < 20 events per hour.

SECONDARY OUTCOMES:
Night 7 responder rate | Night 7
  . Responder rate is based on Sher's Criteria, which are defined as having both a ≥ 50% reduction in AHI and a final AHI of < 20 events per hour.
Night 1 responder rate by baseline disease severity | Night 1
  Responder rate presented by disease severity in accordance with AASM scoring guidelines. Responder rate is based on Sher's Criteria, which are defined as having both a ≥ 50% reduction in AHI and a final AHI of < 20 events per hour.
Night 7 RXiBreeze PAP System compliance rate | Night 7
  Compliance rate is measure of subject use of the RXiBreeze PAP System presented by descriptive statistics.
Nights 1 and 7 Oxygen Desaturation Index (ODI) | Nights 1 and 7
  ODI is average number of desaturation episodes per hour. ODI will be presented by descriptive statistics.
Nights 1 and 7 percentage of time oxygen saturation is < 90% (T90) | Nights 1 and 7
  Oxygen saturation is a measure of the amount of oxygen that is circulating in the blood. T90 oxygen saturation will be presented by descriptive statistics.
Event Detection Validation - Obstructive Apnea Index (OAI) on Night 1 and Night 7 | Nights 1 and 7
  Obstructive Apnea Index (OAI) as measured by the test device (RXiBreeze PAP System) will be compared to the OAI as measured by polysomnography (PSG) to validate accuracy of the test device at nights 1 and 7. Frequency and percentages will be presented.
Event Detection Validation: Hypopnea Index (HI) on Night 1 and Night 7 | Nights 1 and 7
  Event Detection Validation: Hypopnea Index (HI) as measured by the test device (RXiBreeze PAP System) will be compared to the HI as measured by polysomnography (PSG) to validate accuracy of the test device at nights 1 and 7. Frequency and percentages will be presented.
Event Detection Validation: Central Apnea Index (CAI) on Night 1 and Night 7 | Nights 1 and 7
  Event Detection Validation: Central Apnea Index (CAI) as measured by the test device (RXiBreeze PAP System) will be compared to the CAI as measured by polysomnography (PSG) to validate accuracy of the test device at nights 1 and 7. Frequency and percentages will be presented.
Event Detection Validation: Apnea Index (AI) on Night 1 and Night 7 | Nights 1 and 7
  Event Detection Validation: Apnea Index (AI) as measured by the test device (RXiBreeze PAP System) will be compared to the AI as measured by polysomnography (PSG) to validate accuracy of the test device at nights 1 and 7. Frequency and percentages will be presented.
Epworth Sleepiness Scale (ESS) on Night 1 and Night 7 | Nights 1 and 7
  Epworth Sleepiness Scale (ESS) is a validated patient reported outcome (PRO) questionnaire consisting of 8 questions related to daytime sleepiness. The ESS results in a score from 0 to 24 (0 - 10 reflect normal levels of daytime sleepiness, scores over 10 reflect excessive daytime sleepiness (EDS), scores of 16 or more suggest a high level of EDS. The ESS will be self-administered by subjects at the Night 1 and Night 7 visits. Results will be presented by frequency and percentages.
Functional Outcomes of Sleep Questionnaire short form (FOSQ-10) on Night 1 and Night 7 | Nights 1 and 7
  Functional Outcomes of Sleep Questionnaire (FOSQ) short form is a validated patient reported outcome (PRO) questionnaire consisting of 10 questions related to the impact of sleepiness on the ability to conduct daily activities. The FOSQ-10 questions are rates on a scale of 1 to 4 (1=extreme difficulty and 4=no difficulty). A total score and 5 subscale scores (vigilance, general productivity, social outcome, intimacy, and activity level) are calculated. Subscale scores range from 1 (maximum difficulty) to 4 (no difficulty).

OTHER OUTCOMES:
Safety Endpoint: Device- and/or therapy-related adverse events (AEs) | Night 1 through completion of Night 7
  Device- and/or therapy-related adverse events (AEs) will be collected from the Night 1 visit through completion of the Night 7 visit. AEs will be coded using the standardized Medical Dictionary for Regulatory Activities (MedDRA). AEs will be reported by subject and event.

CONTACTS AND LOCATIONS:
Overall Officials: Mehran Farid, MD, Principal Investigator — Peninsula Sleep Center
Locations (9):
- United States (9):
  - Peninsula Sleep Center, Burlingame, California
  - Exalt Clinical Research, Chula Vista, California
  - Bay Sleep Clinic, Mountain View, California
  - Innovative Sleep Centers, Inc., Redding, California
  - TriValley Sleep Center, San Ramon, California
  - NeuroTrials Research, Atlanta, Georgia
  - Somnos Clinical Research, Lincoln, Nebraska
  - Intrepid Research, Cincinnati, Ohio
  - Innovative Sleep Centers, PLLC, Tumwater, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kapur VK, Auckley DH, Chowdhuri S, Kuhlmann DC, Mehra R, Ramar K, Harrod CG. Clinical Practice Guideline for Diagnostic Testing for Adult Obstructive Sleep Apnea: An American Academy of Sleep Medicine Clinical Practice Guideline. J Clin Sleep Med. 2017 Mar 15;13(3):479-504. doi: 10.5664/jcsm.6506. PMID 28162150
- [Background] Sher AE, Schechtman KB, Piccirillo JF. The efficacy of surgical modifications of the upper airway in adults with obstructive sleep apnea syndrome. Sleep. 1996 Feb;19(2):156-77. doi: 10.1093/sleep/19.2.156. PMID 8855039
- [Background] Benjafield AV, Ayas NT, Eastwood PR, Heinzer R, Ip MSM, Morrell MJ, Nunez CM, Patel SR, Penzel T, Pepin JL, Peppard PE, Sinha S, Tufik S, Valentine K, Malhotra A. Estimation of the global prevalence and burden of obstructive sleep apnoea: a literature-based analysis. Lancet Respir Med. 2019 Aug;7(8):687-698. doi: 10.1016/S2213-2600(19)30198-5. Epub 2019 Jul 9. PMID 31300334
- [Background] Kushida CA, Chediak A, Berry RB, Brown LK, Gozal D, Iber C, Parthasarathy S, Quan SF, Rowley JA; Positive Airway Pressure Titration Task Force; American Academy of Sleep Medicine. Clinical guidelines for the manual titration of positive airway pressure in patients with obstructive sleep apnea. J Clin Sleep Med. 2008 Apr 15;4(2):157-71. PMID 18468315